CLINICAL TRIAL: NCT00049738
Title: Screening, Evaluation, Diagnosis, Treatment Optimization and Follow-up for Childhood Onset Psychotic Disorders
Brief Title: Screening for Childhood-Onset Psychotic Disorders
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030035; 03-M-0035
Record Dates: First submitted 2002-11-12; First posted 2002-11-13 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10-05

CONDITIONS: Childhood Onset Psychotic Disorders; Schizophrenia; Psychosis; Psychotic Disorder
Keywords: Psychosis; Childhood Onset Schizophrenia; Schizophrenia; Schizoaffective; Psychotic Disorder; Multidimensionally Impaired Syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to screen and evaluate children with psychotic disorders to establish or confirm their diagnosis and to collect data about their condition. This study will also recruit individuals for various treatment studies.

Childhood psychotic disorders are debilitating conditions in which children have auditory or visual hallucinations and disorganized thoughts. This study will examine psychotic disorders in children in an inpatient setting.

Participants in this study will be admitted to the NIH Clinical Center for up to 9 weeks under one or more of the following conditions: current medication, no medication, or tapered medication. Participants will undergo blood, urine, metabolic, and intellectual functioning tests. An electrocardiogram (EKG) and electroencephalogram (EEG) will be performed. A magnetic resonance imaging (MRI) scan of the brain will be taken and infrared oculography will be used to measure eye movements. Participants and their family members may also be asked to participate in a study of genetics in children with psychotic illnesses. Children meeting criteria for childhood onset schizophrenia may be offered participation in a medication comparison protocol.

DETAILED DESCRIPTION:
Up to 250 children and adolescents ages 5 to 18, meeting DSM IV criteria for schizophrenia, schizoaffective disorder, and psychotic disorder not otherwise specified, are currently under study in our group. The purpose of this protocol is to allow systematic outpatient, and subsequent inpatient, screening evaluation to establish an accurate diagnosis for research, obtain clinical and neurobiological research measurements, evaluate the patient s response to open treatment with antipsychotic(s), and allow longitudinal follow-up. Subjects and first-degree relatives may then be enrolled in Protocol 89-M-0006, Brain Imaging of Childhood Onset Psychiatric Disorders, Endocrine Disorders and Healthy Controls, and Protocol 84-M-0050, Biochemical, Physiological, and Psychological Measures in Normal Controls and Relatives of Psychiatric Patients. If additional research protocols are available, this screening protocol will represent an entry point for them.

The evaluation process will include a one-day outpatient psychiatric screening interview with proband and family. If it is thought that the child is likely to meet criteria for childhood onset psychoses, an inpatient evaluation will then be offered for clarifying the diagnosis. This may involve: 1) Up to 3 weeks of inpatient observation on the child s current medication regimen. 2) Tapering of psychotropic medications (1-4 weeks, depending upon type and dosage). 3) Observation for up to 3 weeks drug free, in order to confirm the diagnosis, and 4) Once the diagnosis is confirmed, two to ten weeks of treatment with antipsychotic(s); 5) Discharge to the care of his/her community psychiatrist. Treatment will be guided by what is considered the subject s best clinical interest. During the inpatient stay, or occasionally as part of the outpatient screening, we will obtain neurocognitive testing, research blood draws including blood for genetic testing of the proband, and a research brain MRI scan. A skin biopsy may be obtained either during the inpatient stay or a follow up visit.

This protocol also includes a study 100 non-schizophrenic children ages 6-13 with psychotic symptoms (e.g. hallucinations or delusions) to extend our studies of early neuro-developmental biomarkers and of the factors that either promote or stop the progression to full schizophrenia (resilience or conversion factors). These children will be recruited from the local community, evaluated as outpatients and followed prospectively for five years. Measures will include diagnostic interviews, clinical ratings, neurocognitive testing, anatomic and functional imaging, and blood for routine and genetic testing.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males and females between the ages of 5 and 18
* Onset of psychotic symptoms before 13th birthday and a presumptive diagnosis of either schizophrenia, schizoaffective disorder, MDI syndrome, or psychosis NOS
* Pre-psychotic IQ 70 or above.

EXCLUSION CRITERIA:

-Major neurological or medical condition (e.g. temporal lobe epilepsy for which patient is on active treatment), or other psychiatric diagnosis that is the main focus of treatment (e.g. serious eating disorder).

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2002-10-29; Study Completion 2017-10-05

PRIMARY OUTCOMES:
Accurate Diagnosis | On going

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Rapoport, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cantor S, Evans J, Pearce J, Pezzot-Pearce T. Childhood schizophrenia: present but not accounted for. Am J Psychiatry. 1982 Jun;139(6):758-62. doi: 10.1176/ajp.139.6.758. PMID 7081488
- [Background] Green WH, Campbell M, Hardesty AS, Grega DM, Padron-Gayol M, Shell J, Erlenmeyer-Kimling L. A comparison of schizophrenic and autistic children. J Am Acad Child Psychiatry. 1984 Jul;23(4):399-409. doi: 10.1016/s0002-7138(09)60317-4. No abstract available. PMID 6747145
- [Background] Beitchman JH. Childhood schizophrenia. A review and comparison with adult-onset schizophrenia. Psychiatr Clin North Am. 1985 Dec;8(4):793-814. PMID 3878510
- [Derived] Markovic A, Buckley A, Driver DI, Dillard-Broadnax D, Gochman PA, Hoedlmoser K, Rapoport JL, Tarokh L. Sleep spindle activity in childhood onset schizophrenia: Diminished and associated with clinical symptoms. Schizophr Res. 2020 Sep;223:327-336. doi: 10.1016/j.schres.2020.08.022. Epub 2020 Sep 24. PMID 32980206
- [Derived] Craddock KES, Zhou X, Liu S, Gochman P, Dickinson D, Rapoport JL. Symptom dimensions and subgroups in childhood-onset schizophrenia. Schizophr Res. 2018 Jul;197:71-77. doi: 10.1016/j.schres.2017.10.045. Epub 2017 Nov 13. PMID 29146021
- [Derived] Kasoff LI, Ahn K, Gochman P, Broadnax DD, Rapoport JL. Strong Treatment Response and High Maintenance Rates of Clozapine in Childhood-Onset Schizophrenia. J Child Adolesc Psychopharmacol. 2016 Jun;26(5):428-35. doi: 10.1089/cap.2015.0103. Epub 2016 Jan 19. PMID 26784704
- [Derived] Berman RA, Gotts SJ, McAdams HM, Greenstein D, Lalonde F, Clasen L, Watsky RE, Shora L, Ordonez AE, Raznahan A, Martin A, Gogtay N, Rapoport J. Disrupted sensorimotor and social-cognitive networks underlie symptoms in childhood-onset schizophrenia. Brain. 2016 Jan;139(Pt 1):276-91. doi: 10.1093/brain/awv306. Epub 2015 Oct 22. PMID 26493637
- [Derived] Anvari AA, Friedman LA, Greenstein D, Gochman P, Gogtay N, Rapoport JL. Hippocampal volume change relates to clinical outcome in childhood-onset schizophrenia. Psychol Med. 2015;45(12):2667-74. doi: 10.1017/S0033291715000677. Epub 2015 May 4. PMID 25936396